CLINICAL TRIAL: NCT01975844
Title: The Effect of Epogen and Venofer Dosing Management on Hemoglobin Stability
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has been terminated due to lack of financial support
Sponsor: Michael Germain (Other)
Collaborators: Western New England Renal & Transplant Associates, PC (Other)
Responsible Party: Sponsor-Investigator, Michael Germain, Medical Director, Renal Transplantation, Department of Medicine, Baystate Medical Center
Organization: Baystate Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-12-197
Record Dates: First submitted 2013-08-13; First posted 2013-11-05 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Anemia; End Stage Renal Disease
Keywords: Anemia; End Stage Renal Disease
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualized Anemia Mangement Protocol (Experimental): Single arm study, therefore all patients will participate in the following:
  Phase 1 (1-3 months): Develop individualized patient models and Anemia Management Protocols (AMP) while patients are receiving standard medical care.
  Phase 2 (9 months): Individualized AMP study period. Phase 3 (9 months): Follow up period: return to standard-care AMP .
  Interventions: Other: Individualized Anemia Mangement Protocol

INTERVENTIONS:
Other: Individualized Anemia Mangement Protocol — Phase 1 (1-3 months): Develop individualized patient models and Anemia Management Protocols (AMP) while patients are receiving standard medical care.
  Phase 2 (9 months): Individualized AMP study period. Phase 3 (9 months): Follow up period: return to standard-care AMP .

SUMMARY:
Hypothesis: Routine clinical tests with feedback control based Epogen(Epo)/Venofer(Iron) protocol will improve Hemoglobin (Hgb) stability and increase the time that patients remain in target

Objectives:

1. Decreased variability of Hgb
2. Increase the % of patients in target range c Increase in time that Hgb remains target range

DETAILED DESCRIPTION:
Study Design One dialysis unit shift comprising up to 200 patients. Study participation will last for 12 months broken into 3 phases as described below.

Phase 1 (1-3 months): Develop individualized patient models and Anemia Management Protocols (AMP) while patients are receiving standard medical care.

Phase 2 (9 months): Individualized AMP study period. Phase 3 (9 months): Follow up period: return to standard-care AMP.

The individual AMP will be utilized weekly during the 9 months of Phase 2.

The 3 objectives will be evaluated and updated weekly, Baseline to Year 1.

All Epo dosing recommendations must be reviewed by the treating physician who can either accept or modify doses at his/her discretion based on clinical event that are not includes in the transmitted data such as bleeding, infection, and hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Receiving hemodialysis in an out-patient dialysis unit

Exclusion Criteria:

* Not receiving EPOGEN as part of their standard medical care
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Intraindividual Hemoglobin (Hgb) variability | Evaluated and updated weekly for 52 weeks
  Change in average intraindividual Hgb variability between control period and treatment periods.

SECONDARY OUTCOMES:
Average hemoglobin levels | Evaluated and updated weekly for 52 weeks
  Change in average Hgb levels between control treatment periods, and change in interindividual Hgb variability between control treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Germain, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Chicopee Dialysis Center, Chicopee, Massachusetts, United States